CLINICAL TRIAL: NCT00632996
Title: Effectiveness of Rehabilitation for Subacromial Impingement Syndrome
Brief Title: Exercise and Manual Therapy for Shoulder Subacromial Impingement Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other); University of North Florida (Other); Arcadia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM10320; Proposal #:PT101875
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder pain; shoulder impingement syndrome; manual therapy; rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Rehabilitation; Physical Therapy Modalities; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Exercise, manual therapy, patient education, posture, home exercise program
  Other Names: Physical Therapy; Manual Therapy

SUMMARY:
The purposes of this study are to:

1. determine if a rehabilitation program that consists of exercise and manual therapy reduces pain and improves quality of life in patients with shoulder subacromial impingement syndrome;
2. determine which patients are likely to respond to this rehabilitation program and which patients are not likely to respond to this rehabilitation program

The hypotheses are:

1. the rehabilitation treatment program will result in significant changes in pain and quality of life
2. there will be items from the history and examination that will identify those patients who respond favorably and those who do not respond favorably to rehabilitation at 6 weeks, 3, 6 and 12 months.

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SAIS) is the most frequent cause of shoulder pain. A variety of non-surgical treatments have been advocated to correct the impairments associated with SAIS. Clinical trials support the use of therapeutic exercise and joint mobilizations to improve pain and functional disability associated with SAIS. However, not all patients in these trials had a favorable outcome. Moreover, the effect sizes in these trials were small to moderate. Thus the purposes of this study are to 1. determine the effect of a multi-modal rehabilitation program consisting of strengthening, stretching, manual therapy to the shoulder and spine, patient education, posture, and functional re-training; and 2. identify those patients who are and who are not likely to respond to rehabilitation at the start of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of shoulder impingement syndrome as evidence by all 5 criteria:

  1. Reproduction of symptoms with impingement test: either Hawkins-Kennedy or Neer Test
  2. Pain during active shoulder elevation at or above 60 degrees
  3. Weakness of rotator cuff or pain during the Empty Can test or during resisted shoulder external rotation
  4. Shoulder disability: greater than or equal to 20/100 (0 = no disability)
  5. Able to understand written and spoken English

Exclusion Criteria:

* Severe pain; pain is > or equal to 7/10 on NPRS (0 = no pain)
* Shoulder surgery on affected shoulder
* Traumatic shoulder dislocation within the past 3 months
* Previous rehabilitation for this episode of shoulder pain
* Reproduction of shoulder pain with active or passive cervical motion
* Systemic inflammatory joint disease
* Global loss of passive shoulder ROM, indicative of adhesive capsulitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Shoulder disability | 6 week and 3, 6, 12 months

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks and 3, 6, 12 months
Quality of life | 6 weeks and 3, 6, 12 months
Pain with rest, normal activities, and strenuous activities | 6 weeks and 3, 6, 12 months
Patient perceived global rating of effect | 6 weeks and 3 months
Additional healthcare utilization and medication use | 6 weeks and 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Michener, PhD, PT, ATC, Principal Investigator — Virginia Commonwealth University; Phillip W McClure, PhD, PT, Principal Investigator — Arcadia University; Angela R Tate, PhD, PT, Study Director — Arcadia University; Ian A Young, PT, Study Chair — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Tate AR, McClure PW, Young IA, Salvatori R, Michener LA. Comprehensive impairment-based exercise and manual therapy intervention for patients with subacromial impingement syndrome: a case series. J Orthop Sports Phys Ther. 2010 Aug;40(8):474-93. doi: 10.2519/jospt.2010.3223. PMID 20710088